CLINICAL TRIAL: NCT06620003
Title: A Phase 2, Randomized, Double-blind, Placebo-Controlled Trial to Evaluate Safety, Tolerability, and Immune Responses of an Investigational Monovalent Chimpanzee Adenoviral Vectored Marburg Virus Vaccine in Healthy Adults
Brief Title: A Trial to Evaluate Safety, Tolerability, and Immune Responses of an Investigational Monovalent Chimpanzee Adenoviral Vectored Marburg Virus Vaccine in Healthy Adults
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Albert B. Sabin Vaccine Institute (Other)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Sabin-004; 75A05119C00055 (Other Grant/Funding Number: DHHS/ASPR-BARDA)
Record Dates: First submitted 2024-09-18; First posted 2024-10-01 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Marburg Virus Disease
Keywords: Marburg Virus; Marburg Vaccine; cAd3-Marburg vaccine
MeSH Terms: conditions — Marburg Virus Disease

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 4:1 to receive the cAd3-Marburg Vaccine at 1.0 × 10^11 PU/dose or placebo (normal saline; 0.9% sodium chloride (NaCl) solution for injection) at Day 1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- cAd3-Marburg Vaccine (1.0 × 10^11 PU) (Active Comparator): Single dose of cAd3-Marburg Vaccine (1x10^11 PU) administered intramuscularly (IM) with needle and syringe in a volume of 0.71 mL.
  Interventions: Biological: cAd3-Marburg Vaccine
- Placebo 0.9% NaCl solution (Placebo Comparator): Single dose of Placebo (0.9% NaCl solution for injection) administered intramuscularly (IM) with needle and syringe in a volume of 0.71 mL.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: cAd3-Marburg Vaccine — The recombinant chimpanzee adenovirus Type 3-vectored Marburg vaccine, (cAd3-Marburg Vaccine) is composed of a cAd3 vector that expresses Marburg wild type glycoprotein (WT GP) from the Angola strain.
  Arms: cAd3-Marburg Vaccine (1.0 × 10^11 PU)
Biological: Placebo — 0.9% NaCl solution for injection.
  Arms: Placebo 0.9% NaCl solution

SUMMARY:
A Phase 2, Randomized, Double-blind, Placebo-Controlled Trial to Evaluate Safety, Tolerability, and Immune Responses of an Investigational Monovalent Chimpanzee Adenoviral Vectored Marburg Virus Vaccine in Healthy Adults

DETAILED DESCRIPTION:
This is a multi-center, double-blinded, placebo-controlled, Phase 2 study to evaluate safety, tolerability, and immunogenicity of a single dose of cAd3-Marburg Vaccine in healthy adults 18 to 70 years of age, in a US-based population. The study will enroll 200 eligible participants randomized 4:1 to receive the cAd3-Marburg Vaccine at 1.0 × 10^11 PU/dose or placebo (normal saline; 0.9% sodium chloride (NaCl) solution for injection) at Day 1, intramuscularly, in deltoid muscle. Participants will be screened for eligibility up to 28 days before enrollment. Safety data will be periodically reviewed by an independent DSMB. Safety and immunogenicity will be assessed at Days 1, 8, 15, 29, 85, 169, and will conclude at the end of study visit on Day 366. PBMCs will be collected from a subset of 40 subjects on days 1, 15, 29, 169 and will conclude at the end of study visit on Day366 to access cellular immunity. All participants will also be contacted telephonically on Days 4 and 42 (unless a clinic visit is medically indicated, or participant does not have a phone contact) for safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to complete and provide informed consent prior to any trial procedure including optional consent for retention of blood samples for potential future testing and assay development. As part of the informed consent process, the participant must complete a Test of Understanding (ToU) about the study and answer at least 90% of the questions correctly at least once in three attempts.
2. Male or non-pregnant female 18 to 70 (inclusive) years of age at time of consent;
3. Is capable of understanding and agrees to comply with planned trial procedures and to be available for all clinic follow-up for all planned trial visits;
4. Able to provide proof of identity to the satisfaction of the trial clinician completing the enrollment process; has a means to be contacted and to contact the investigator during the trial;
5. Agree not to receive any vaccine within 3 months of trial vaccination (prior and after) trial;
6. Agree not to donate bone marrow, blood, or blood products until 3 months after the trial vaccination;
7. In good general health without clinically significant medical conditions, based on medical history, physical examination, vital signs, and clinical laboratory results as deemed acceptable by PI;
8. Clinical laboratory results within 28 days prior to vaccination within the testing laboratory reference ranges (or deemed not clinically significant by the PI) for the following parameters: White blood cells (WBC), Complete blood count (CBC), Red blood cells (RBC), Hemoglobin (HGB), total lymphocyte count, coagulation tests to include prothrombin time in terms of INR, fibrinogen, protein C, d-dimer, and chemistry tests to include alanine aminotransferase (ALT), aspartate aminotransferase (AST), and serum creatinine. A laboratory result that is outside the reference range and is deemed not clinically significant by the PI will not exclude the participant;
9. Has a body mass index (BMI) > 17 and ≤ 37 at screening.

   Female participant specific criteria:
10. Negative pregnancy serum test at screening, and negative urine pregnancy test before vaccination AND:
11. Use of oral, implantable, transdermal or injectable contraceptives for 21 days prior to vaccination and for at least 24 weeks after vaccination, UNLESS the female participant fulfills one of the following criteria:

    1. At least 1 year post-menopausal.
    2. Surgically sterile.
    3. Use of another reliable form of contraception must be approved by the Investigator (e.g., double barrier method, intrauterine device, contraceptive patches).

    Male participants must agree:
12. Not to father a child or donate sperm for at least 24 weeks after vaccination;
13. To use an effective means of birth control from at least 21 days prior to vaccination and for at least 24 weeks after vaccination if assessed to be of reproductive potential.

Exclusion Criteria:

1. Participant is female and is breastfeeding or plans to become pregnant or breastfeed from trial vaccination through 24 weeks post-vaccination
2. Has any medical disease or condition that, in the opinion of the investigator, precludes trial participation. This includes any acute, subacute, intermittent, or chronic medical disease or condition that would place the Participant at an unacceptable risk of injury, render the Participant unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the Participant's successful completion of the trial; (Chronic conditions that are well-controlled and medically stable, i.e. no relevant change in treatment for medical reasons occurred in the last 6 months, are allowed at the discretion of the PI, e.g. hypertension, asthma, thyroid disease) Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g., malignancy, Human Immunodeficiency Virus [HIV] infection) or immunosuppressive/cytotoxic therapy (e.g., medications used during cancer chemotherapy, organ transplantation or to treat autoimmune disorders) and any infection requiring IV antibiotics or hospitalization within 90 days prior to screening
3. History of Guillain-Barré syndrome
4. History of allergy to any component of the vaccine
5. Serology screen positive for infectious diseases (hepatitis B, hepatitis C, HIV, Human T-cell leukemia virus (HTLV), Syphilis);
6. Known prior exposure to Marburg virus or prior diagnosis of Marburg Virus Disease, determined from the participant's reported medical history
7. History of or active status of any of the following clinically significant conditions:

   1. Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain;
   2. Allergic reaction to excipients in the trial vaccine including gentamycin, neomycin or streptomycin;
   3. Diabetes mellitus Type I or Type II (even if stable)
   4. Tuberculosis
   5. Hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema;
   6. Idiopathic urticaria within the last year
   7. Any malignancy, including non-skin melanoma, that has been active or treated, within 5 years prior to screening. (If diagnosed malignancy is 5 or more years prior to enrollment and cured with no ongoing treatment the malignancy will NOT be considered an exclusion);
   8. Seizure in the past 3 years or treatment for seizure disorder in the past 3 years (even if stable);
   9. Asplenia or functional asplenia;
   10. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a participant's ability to give informed consent;
8. Hematologic History:

   1. Bleeding disorder diagnosed by a doctor or use of anticoagulant medications such as, Warfarin, Apixaban, Dabigatran (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws;
   2. Family and personal history of bleeding or thrombosis or heparin-induced thrombocytopenia
   3. Conditions known to increase risk of thrombosis (e.g., pregnant or post-partum, extreme obesity, active malignancy or post-transplantation, recent surgery, immobility, recent infection, recent head trauma, autoimmune disease, inflammatory disease),
   4. Receipt of blood products within 3 months prior to enrollment.
   5. Has donated ≥ 450 mL of blood products within 30 days prior to randomization or expects to donate blood within 90 days of vaccine administration
   6. History of heparin-related thrombotic events, and/or receiving heparin treatments
9. Has a clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature ≥38.0° Celsius (≥100.4° Fahrenheit) within 24 hours of the planned dose of trial vaccine, rescreening and randomization at a later date is permitted at the discretion of the investigator and after consultation with the sponsor
10. Receipt of any of the following substances:

    1. prior receipt of Sudan Virus Vaccine or Marburg Vaccine
    2. prior receipt of any adenoviral vectored vaccine, adenovirus-based or adeno-associated virus (AAV)-based gene therapies or treatments, including adenoviral COVID-19 vaccines or boosters.
    3. Participant received an investigational drug (including investigational drugs for prophylaxis of COVID-19) within 3 months of dosing, or has used an invasive investigational medical device within 3 months of dosing
    4. received immunoglobulin (Ig) or monoclonal antibodies within 3 months,
    5. is currently enrolled or plans to participate in another investigational or interventional trial during the course of this trial (observational/registry trials are allowed)
11. Use of systemic corticosteroids in daily dose equivalence > 20 mg of prednisolone in the last 90 days, and for periods exceeding 10 days. Non-steroidal anti-inflammatory drugs [NSAIDS] are permitted.
12. Current anti-tuberculosis prophylaxis or therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of cAd3-Marburg Vaccine, by count and percentage of vaccinated participants who develop: SAEs, solicited/unsolicited AEs, AESI, MAAE, and AE at each intensity level of cAd3-Marburg Vaccine | 1 Year
  Count and percentage of vaccinated participants who develop: serious adverse events (SAEs), solicited adverse events (AEs), unsolicited AEs, adverse event of special interest (AESI), medically attended adverse events (MAAE), and AE at each intensity level. Estimand 1a (Primary): Count and percentage of vaccinated participants who would develop SAEs, solicited AEs, unsolicited AEs, AESI, MAAE, and AE at each intensity level will be evaluated with each treatment group. A treatment policy strategy is used for assessing safety irrespective of a current (or prior) infection at time of the vaccination. Infections and death (if vaccinated participants meet the AE and time window criteria) are included in the endpoint (composite strategy).

SECONDARY OUTCOMES:
To determine the geometric mean concentration (GMC) of anti-Marburg-GP binding IgG antibodies to cAd3-Marburg Vaccine at Day 29 post-vaccination. | 29 Days
  Secondary Endpoint: To evaluate the humoral immunogenicity induced by cAd3-Marburg Vaccine at Day 29 post-vaccination. Estimand 2a: Geometric mean concentration (GMC) of cAd3-Marburg Vaccine will be compared to placebo on Day 29 post-vaccination. The hypothetical strategy is used to estimate antibody levels without subsequent Marburg virus (MARV) infection or influence from immune-modifying drugs or non-trial interventions. The principal stratum strategy excludes those with active or prior MARV infection at the time of the vaccination.
To determine geometric mean increase (GMI) of anti-Marburg-GP binding IgG antibodies at Day 29 post-vaccination | 29 Days
  Secondary Endpoint: To evaluate the humoral immunogenicity induced by cAd3-Marburg Vaccine at Day 29 post-vaccination. Estimand 2b: Geometric mean increase (GMI) of anti-Marburg-GP binding IgG antibodies against Marburg-GP on Day 29. The hypothetical strategy is used to estimate antibody levels without subsequent Marburg virus (MARV) infection or influence from immune-modifying drugs or non-trial interventions. The principal stratum strategy excludes those with active or prior MARV infection at the time of the vaccination.
To determine the geometric mean of the ND50 (GMND50) of anti-Marburg-GP neutralizing antibodies on Day 29 post-vaccination. | 29 Days
  Secondary Endpoint: To evaluate the humoral immunogenicity induced by cAd3-Marburg Vaccine at Day 29 post-vaccination. Estimand 2c: The geometric mean of the ND50 (GMND50) of anti-Marburg-GP neutralizing antibodies on Day 29. The hypothetical strategy is used to estimate antibody levels without subsequent Marburg virus (MARV) infection or influence from immune-modifying drugs or non-trial interventions. The principal stratum strategy excludes those with active or prior MARV infection at the time of the vaccination.
To determine the geometric mean increase of the ND50 (GMIND50) of anti-Marburg-GP neutralizing antibodies at Day 29 post-vaccination. | 29 Days
  Secondary Endpoint: To evaluate the humoral immunogenicity induced by cAd3-Marburg Vaccine at Day 29 post-vaccination. Estimand 2d: The geometric mean increase of the ND50 (GMND50) of anti-Marburg-GP neutralizing antibodies on Day 29. The hypothetical strategy is used to estimate antibody levels without subsequent Marburg virus (MARV) infection or influence from immune-modifying drugs or non-trial interventions. The principal stratum strategy excludes those with active or prior MARV infection at the time of the vaccination.
To determine the percentage of participants (and 95%CI) with seroconversion at Day 29 post-vaccination. | 29 Days
  Secondary Endpoint: To evaluate the humoral immunogenicity induced by cAd3-Marburg Vaccine at Day 29 post-vaccination. Estimand 2e: Percentage of participants (and 95%CI) with seroconversion at Day 29. The hypothetical strategy is used to estimate antibody levels without subsequent Marburg virus (MARV) infection or influence from immune-modifying drugs or non-trial interventions. The principal stratum strategy excludes those with active or prior MARV infection at the time of the vaccination.
To determine the geometric mean concentration (GMC) of anti-Marburg-GP binding IgG antibodies on Day 1, Day 8, Day 15, Day 85, Day 169, and Day 366. | 1 Year
  Secondary Endpoint: To evaluate the humoral immunogenicity induced by cAd3-Marburg Vaccine across additional trial timepoints. Estimand 3a: GMCs of anti-Marburg-GP binding IgG antibodies on Day 1, Day 8, Day 15, Day 85, Day 169, and Day 366. The hypothetical strategy is used to estimate antibody levels without subsequent Marburg virus (MARV) infection or influence from immune-modifying drugs or non-trial interventions. The principal stratum strategy excludes those with active or prior MARV infection at the time of the trial intervention.
To determine the geometric mean increase (GMI) of anti-Marburg-GP binding IgG antibodies against Marburg-GP at optional selected timepoints (Day 8, Day 15, Day 85, Day 169, and Day 366). | 1 Year
  Secondary Endpoint: To evaluate the humoral immunogenicity induced by cAd3-Marburg Vaccine across additional trial timepoints. Estimand 3b: GMI of anti-Marburg-GP binding IgG antibodies against Marburg-GP at optional selected timepoints (Day 8, Day 15, Day 85, Day 169, and Day 366). The hypothetical strategy is used to estimate antibody levels without subsequent Marburg virus (MARV) infection or influence from immune-modifying drugs or non-trial intervention. The principal stratum strategy excludes those with active or prior MARV infection at the time of the trial intervention.
To determine geometric mean increase of the ND50 (GMIND50) of anti-Marburg-GP neutralizing antibodies on Day 1, Day 8, Day 15, Day 85, Day 169, and Day 366. | 1 Year
  Secondary Endpoint: To evaluate the humoral immunogenicity induced by cAd3-Marburg Vaccine across additional trial timepoints. Estimand 3c: GMIND50 of anti-Marburg-GP neutralizing antibodies on Day 1, Day 8, Day 15, Day 85, Day 169, and Day 366. The hypothetical strategy is used to estimate antibody levels without subsequent Marburg virus (MARV) infection or influence from immune-modifying drugs or non-trial interventions. The principal stratum strategy excludes those with active or prior MARV infection at the time of the trial intervention.
To determine geometric mean increase of ND50 of anti-Marburg-GP neutralizing antibodies at optionally selected timepoints (Day 8, Day 15, Day 85, Day 169, and Day 366) | 1 Year
  Secondary Endpoint: To evaluate the humoral immunogenicity induced by cAd3-Marburg Vaccine across additional trial timepoints. Estimand 3d: GMIND50 of anti-Marburg-GP neutralizing antibodies at optionally selected timepoints (Day 8, Day 15, Day 85, Day 169, and Day 366). The hypothetical strategy is used to estimate antibody levels without subsequent Marburg virus (MARV) infection or influence from immune-modifying drugs or non-trial interventions. The principal stratum strategy excludes those with active or prior MARV infection at the time of the trial intervention.
To determine the percentage of participants (and 95%CI) with seroconversion at Day 8, Day 15, Day 85, Day 169, and Day 366. | 1 Year
  Secondary Endpoint: To evaluate the humoral immunogenicity induced by cAd3-Marburg Vaccine across additional trial timepoints. Estimand 3e: Percentage of Participants (and 95%CI) with seroconversion at Day 8, Day 15, Day 85, Day 169, and Day 366. The hypothetical strategy is used to estimate antibody levels without subsequent Marburg virus (MARV) infection or influence from immune-modifying drugs or non-trial interventions. The principal stratum strategy excludes those with active or prior MARV infection at the time of the trial intervention.

OTHER OUTCOMES:
To determine cell-mediated immune response to cAd3-Marburg Vaccine at Day 1, Day 15, Day 29, Day 169, and Day 366 in a subset of 40 Participants | 1 Year
  Exploratory Objective: If deemed necessary, to further characterize the immune response of cAd3-Marburg Vaccine. Estimand 4a: Frequency of IFN-γ secreting T-cells by ELISpot. Percentage of CD4+ T-cells and/or CD8+ T-cells that producing IFN-γ and/or IL-2 and/or TNF-α, as measured by ICS.
To determine the geometric mean concentration (GMC) of anti-Marburg-GP binding IgM antibodies at Day 1, Day 8, Day 15, and Day 29. | 29 Days
  Exploratory Objective: If deemed necessary, to further characterize the immune response of cAd3-Marburg Vaccine. Further exploratory immunology to detect cAd3-Marburg Vaccine-related immune responses. Estimand 4b: The GMC of anti-Marburg-GP binding IgM antibodies at Day 1, Day 8, Day 15, and Day 29.
To determine Systems serology (multiple assays in high throughout screen) D1 and D29 | 29 Days
  Exploratory Objective: If deemed necessary, to further characterize the immune response of cAd3-Marburg Vaccine. Further exploratory immunology to detect cAd3-Marburg Vaccine-related immune responses. Estimand 4c: Systems serology (multiple assays in high throughout screen) D1 and D29

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Optimal Research; LLC, Huntsville, Alabama
  - Synexus Clinical Research US, Inc., Phoenix, Arizona
  - Optimal Research; LLC, Melbourne, Florida
  - Synexus Clinical Research US, Inc., Chicago, Illinois
  - Optimal Research; LLC, Peoria, Illinois
  - Synexus Clinical Research US; Inc., Dallas, Texas
  - Synexus Clinical Research US, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The clinical trial results will be published in a peer-reviewed journal, which will include, as feasible, the study protocol. A summary of the study results will be included within the trial registration records in ClinicalTrials.gov.
Time Frame: The sponsor will also publish results in a manuscript in a peer reviewed journal, which requires a published study protocol. The sponsor expects this will be done by early 2027.